CLINICAL TRIAL: NCT00274781
Title: A Phase II Trial of Combination Therapy With Arsenic Trioxide (Trisenox) and Gemtuzumab Ozogamicin (Mylotarg) for the Treatment of Adult Patients With Advanced Myelodysplastic Syndrome
Brief Title: Arsenic Trioxide and Gemtuzumab Ozogamicin in Treating Patients With Advanced Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of Michigan (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF6818; P30CA043703 (NIH); CCF-6818 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; chronic myelomonocytic leukemia; secondary acute myeloid leukemia; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; de novo myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Arsenic Trioxide; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATO + GO (Experimental): Arsenic Trioxide 0.25 mg/kg D1-5 Week 1/Twice Weekly W2-12 + Gemtuzumab Ozogamicin 3 mg/m^2 D8 for 1 or 2 Cycles of 12 Weeks each
  Interventions: Drug: arsenic trioxide; Drug: gemtuzumab ozogamicin

INTERVENTIONS:
Drug: arsenic trioxide — Arsenic trioxide will be administered at a dose of 0.25 mg/kg/day IV over 1-2 hours for 5 consecutive days during the first week. Subsequently, arsenic trioxide will be given at a dose of 0.25mg/kg/day twice a week for 11 additional weeks (weeks 2-12).
  Other Names: Trisenox
Drug: gemtuzumab ozogamicin — Gemtuzumab ozogamicin consists of a 2 hr infusion at a dose of 3mg/m2 on day 8 of each 12-week cycle. Gemtuzumab ozogamicin should be administered at a minimum of one hour after the completion of the arsenic trioxide infusion
  Other Names: Mylotarg

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide and gemtuzumab ozogamicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving arsenic trioxide together with gemtuzumab ozogamicin works in treating patients with advanced myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of arsenic trioxide and gemtuzumab ozogamicin to achieve complete and partial remissions in patients with advanced myelodysplastic syndromes.

Secondary

* Determine the efficacy of this regimen, in terms of 50% decrease in Red Blood Cell (RBC) transfusion requirements and change in hemoglobin concentration from baseline in patients treated with this regimen.
* Determine the platelet, neutrophil, bone marrow, and cytogenic response in patients treated with this regimen.
* Determine the response duration in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the safety and toxicity of this regimen in these patients.

OUTLINE: This is a multicenter, open-label study.

Patients receive arsenic trioxide IV over 1 hour once daily on days 1-5 in week 1 and then twice weekly in weeks 2-12. They also receive gemtuzumab ozogamicin IV over 2 hours on day 8. Treatment repeats every 12 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 12 weeks during study treatment, and then 4 weeks after the completion of study treatment.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following hematologic malignancies:

  * Myelodysplastic syndromes (MDS) of one of the following French-American-British (FAB) classifications:

    * Refractory anemia with excess blasts (RAEB) (WHO RAEB-1)
    * RAEB in transformation (RAEB-t) (RAEB-2)
    * Chronic myelomonocytic leukemia (CMML) with > 5% myeloblasts (WHO CMML-2)
  * International Prognostic Scoring System (IPSS) score of intermediate-2 or higher in the setting of > 5% myeloblasts
  * Acute myeloid leukemia that has evolved from MDS
* Must not be a candidate for bone marrow transplantation as first-line therapy or must have declined bone marrow transplantation

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of at least 4 months
* Serum potassium ≥ 4.0 milliequivalent (mEq/dL) and serum magnesium ≥ 1.8 mg/dL (supplemental electrolytes allowed)
* Absolute corrected QT interval (QTc) interval < 460 msec
* No serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the patient at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent
* Not pregnant or nursing
* Fertile patients must be willing to use adequate contraception (barrier method with spermicidal jelly, intrauterine device (IUD), or oral contraceptives)
* Negative pregnancy test
* Creatinine > 2.5 mg/dL
* serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) > 1.5 times upper limit of normal
* Bilirubin > 2.0 mg/dL
* No history of malignancy within the past 3 years other than MDS except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* Arsenic trioxide is contraindicated in patients who are hypersensitive to arsenic

PRIOR CONCURRENT THERAPY:

* No prior bone marrow transplantation
* Must not receive another investigational or approved therapy for MDS within 4 weeks of study enrollment, including growth factors (within 1 week of study enrollment)
* No prior arsenic trioxide or gemtuzumab ozogamicin
* No other concurrent cytotoxic drugs or investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-02; Primary Completion 2008-12 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikkael A. Sekeres, MD, MS, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at Cleveland Clinic and the University of Michigan from February 2004 through June 2006.
Groups:
- ATO (0.25mg/kg) and GO (3mg/m2): ATO dosing was based on the phase 2 European Union regimen at a dose of 0.25 mg/kg administered intravenously on Days 1 through 5 during Week 1 and then twice weekly during Weeks 2 to 12, and GO at a dose of 3mg/m2 on Day 8 for 1 or 2 cycles of 12 weeks each.
Period: Overall Study
Arm/Group | ATO (0.25mg/kg) and GO (3mg/m2)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ATO (0.25mg/kg) and GO (3mg/m2)
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 69 [44 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Complete and Partial Remission Per the International Working Group (IWG) Criteria for Myelodysplastic Syndromes (MDS) or Acute Myeloid Leukemia (AML)
Description: The null hypothesis to be tested was the percentage who will respond to combination arsenic trioxide (ATO) and gemtuzumab ozogamicin (GO) therapy is <10%. A total of >/= 9 responses observed in 30 evaluable patients was taken as evidence warranting further study of the regimen, provided the toxicity profile also appears favorable. The IWG Criteria standardizes the clinical responses in MDS and AML based upon hematologic improvement, quality of life and cytogenic improvement. These standardizations allow for the responses to be determined as either complete responses or partial responses.
Time Frame: at 12 weeks post treatment
Population: Responses According to IWG MDS Criteria (n=30) Responses According to IWG AML Criteria (n=12)
Measure: Number; unit: percentage of patients
Arm/Group | ATO + GO
Number analyzed (Participants) | 30
percentage of patients
  Responses according to IWG MDS Criteria | 30
  Responses according to IWG AML Criteria | 25
  Responses according to Both Criteria | 10

2. Secondary Outcome: Overall Survival
Description: Patient's Overall Survival from date of enrollment to a minimum of three years for survival.
Time Frame: From date of enrollment to a minimum of three years for survival
Measure: Median (Full Range); unit: months
Arm/Group | ATO (0.25mg/kg) and GO (3mg/m2)
Number analyzed (Participants) | 30
months
  Overall Survival | 9.7 [.75 to 38]
  Responders Overall Survival | 28.6 [3.5 to 38]
  Nonresponders Overall Survival | 7.6 [0.75 to 38]

3. Secondary Outcome: Tolerability
Description: Tolerability of Therapy was assessed through use of the National Cancer Institute Common Toxicity Criteria (version 3.0). Treatment tolerability was determined based upon whether or not the physician determined therapy was in the patient's best interest, whether the patient wanted to continue therapy or not, whether patients discontinued treatment due to progressive disease, or whether patients discontinued treatment due to toxicity.
Time Frame: 12 Weeks
Measure: Number; unit: participants
Arm/Group | ATO (0.25mg/kg) and GO (3mg/m2)
Number analyzed (Participants) | 30
participants
  Patients Who Completed 1 12-Week Cycle (C1) | 17
  Patients Who Completed 2 12-Week Cycles (C2) | 7
  Discontinue Tx During C1: Patient/Physician Choice | 5
  Discontinue Tx During C1: Progressive Disease | 5
  Discontinue Tx During C1:Treatment Toxicity | 3
  Discontinue Tx After C1: Progressive Disease | 8
  Discontinue Tx After C1: Treatment Toxicity | 2

ADVERSE EVENTS:
Time Frame: 12 Weeks of Therapy
Arm/Group | ATO (0.25mg/kg) and GO (3mg/m2)
Serious Adverse Events (participants affected / at risk) | 19/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATO (0.25mg/kg) and GO (3mg/m2) (N=30)
Thrombocytopenia (Vascular disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 19
Anemia (Blood and lymphatic system disorders) | 11
Fatigue (Musculoskeletal and connective tissue disorders) | 4
Nausea / Vomiting / Dyspepsia (Gastrointestinal disorders) | 1
Diarrhea / Constipation (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia (Infections and infestations) | 5
QT / QTc Interval Prolongation (Cardiac disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATO (0.25mg/kg) and GO (3mg/m2) (N=30)
Thrombocytopenia (Vascular disorders) | 16
Neutropenia (Blood and lymphatic system disorders) | 20
Anemia (Blood and lymphatic system disorders) | 22
Fatigue (Musculoskeletal and connective tissue disorders) | 28
Rash / Pruritis (Skin and subcutaneous tissue disorders) | 12
Pain (Musculoskeletal and connective tissue disorders) | 16
Edema (Blood and lymphatic system disorders) | 9
Nausea / Vomiting / Dyspepsia (Gastrointestinal disorders) | 18
Diarrhea / Constipation (Gastrointestinal disorders) | 20
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Anorexia / Decreased Appetite (Metabolism and nutrition disorders) | 10
Pyrexia (Immune system disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Insomnia (General disorders) | 4
Catheter / Infusion Site Disorders / Infections (Infections and infestations) | 4
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 6
Cardiac Arrhythmia (Cardiac disorders) | 8
Pneumonia (Infections and infestations) | 8
Headache (Nervous system disorders) | 11
QT / QTc Interval Prolongation (Cardiac disorders) | 4
Chills / Rigors (Immune system disorders) | 16
Dizziness / Vertigo (Nervous system disorders) | 6
Ecchymosis / Petechiae (Blood and lymphatic system disorders) | 5
Neuropathy (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No